CLINICAL TRIAL: NCT07289958
Title: Effects of Respiratory Muscle Training on Cardiovascular, Respiratory, Metabolic and Physical Exercise Capacity Parameters Related to Obesity in Post-bariatric Surgery Patients
Brief Title: Effects of Respiratory Muscle Training in Post-bariatric Surgery Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ramon Llull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-IMTObes
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery
Keywords: Bariatric Surgery; Inspiratory muscle training; Therapeutic exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The randomization system will be carried out by a researcher who is not involved in the evaluation, intervention and data analysis. This researcher will be responsible for providing the respiratory muscle training devices for the different subject groups, delivering them in opaque envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Sham Comparator): The control group will perform inspiratory muscle training with a simulated device 5 times a week for 12 weeks and usual care.
  Interventions: Other: simulated inspiratory muscle
- Inspiratory muscle training (Experimental): Inspiratory muscle training with intensities of 30% to 60% of maximum inspiratory performing 30 repetitions 5 times a week for 12 weeks and usual care.
  Interventions: Behavioral: Inspiratory muscle training
- Institutionalized therapeutic exercise + simulated inspiratory muscle training (Experimental): Aerobic training with intensities of 50 to 65% of the Reserve Heart Rate, neuromuscular training with intensities of 40 to 70% of 1RM and Inspiratory muscle training with simulated inspiratory muscle training, 5 times a week for 12 weeks.
  Interventions: Behavioral: Inspiratory muscle training; Other: simulated inspiratory muscle
- Institutionalized therapeutic exercise + inspiratory muscle training (Experimental): Aerobic training with intensities of 50 to 65% of the Reserve Heart Rate, neuromuscular training with intensities of 40 to 70% of 1RM and Inspiratory muscle training with intensities of 30% to 60% of maximum inspiratory pressure performing 30 repetitions, 5 times a week for 12 weeks.
  Interventions: Behavioral: Institutionalized therapeutic exercise; Behavioral: Inspiratory muscle training

INTERVENTIONS:
Behavioral: Institutionalized therapeutic exercise — Physical exercise program for cardiometabolic rehabilitation (institutionalized) with aerobic training starting with intensities of 50% to 54% of Heart Rate Reserve from week 1 to 4, increasing from 54% to 60% from week 5 to 8 and from 60% to 65% from week 9 to 12, with volumes of 10 minutes the first week and 20 minutes from week 2 to 12, neuromuscular training with intensities of 40% to 70% of 1RM estimated by OMNI RES scale with volumes of 10 to 15 repetitions 3 to 4 sets, 3 times per week.
  Arms: Institutionalized therapeutic exercise + inspiratory muscle training
Behavioral: Inspiratory muscle training — Inspiratory muscle training using a pressure threshold system exerciser with an initial intensity of 30% of maximum inspiratory pressure, increasing the pressure by 10% every 2 weeks until reaching 60% with a volume of 3 sets of 10 repetitions, 5 times per week for 12 weeks.
  Arms: Inspiratory muscle training; Institutionalized therapeutic exercise + inspiratory muscle training; Institutionalized therapeutic exercise + simulated inspiratory muscle training
Other: simulated inspiratory muscle — Inspiratory muscle training with sham device, 5 times a week for 12 weeks.
  Arms: Control Group; Institutionalized therapeutic exercise + simulated inspiratory muscle training

SUMMARY:
Obesity is a health condition caused by excessive accumulation of body fat. This condition is linked to the development of chronic diseases and also places increased stress on the respiratory system, leading to respiratory disorders, exacerbation of preexisting respiratory conditions, and a decline in physical capacity and exercise tolerance.

Respiratory muscle training has been shown to have beneficial effects on respiratory function in these patients, although the effects this strategy has on other metabolic and physiological aspects related to exercise and obesity that are affected remain unclear.

DETAILED DESCRIPTION:
The present study describes a randomized clinical trial developed for 12 weeks with the purpose of the study is to determine that respiratory muscle training produces positive effects on cardiovascular, respiratory, metabolic and physical exercise capacity parameters related to obesity in post-bariatric surgery patients.

The study divides the subjects into two research arms in a relationship of 2 groups per branch: A) Intervention group: institutionalized therapeutic exercise + inspiratory muscle training device versus control group: institutionalized therapeutic exercise + sham device B) Intervention group: inspiratory muscle training device versus control group: sham device, this to determine how the inspiratory muscle training impacts in combination with physical exercise or in isolation versus physical exercise or usual care.

The evaluation criteria are maximum inspiratory pressure, sleep apnea index, sleep quality, resting heart rate, blood pressure, functional capacity, glycosated hemoglobin, lipid profile, body composition and Health-Related Quality of Life; Assessments will be conducted before and after the 12-week program.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with obesity within 1 month of bariatric surgery
* Both sexes
* Ages 18 to 60

Exclusion Criteria:

* Patients with respiratory conditions that contraindicate physical exercise
* Patients with diagnosed heart disease
* Patients with psychiatric conditions
* Patients with osteoarticular conditions that make physical exercise difficult

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum inspiratory pressure (MIP) | Before and after intervention (12 weeks)
  Maximum inspiratory pressure (MIP) is the maximum level of pressure applied to the lungs during inhalation. In normal breathing, this value reflects a negative pressure in centimeters of water (cm H₂O).
Sleep Apnea | Before and after intervention (12 weeks)
  Sleep apnea is a potentially serious sleep disorder in which breathing stops and starts repeatedly. They are measured with sleep tests that measure heart rate, oxygen levels, airflow, and breathing patterns. The Apnea-Hypopnea Index (AHI) is a measure of the number of times a person stops breathing (apnea) or has shallow breathing (hypopnea) per hour of sleep. A higher AHI indicates greater severity, with typical ranges classifying the condition as mild (5-15 events/hour), moderate (16-30 events/hour), or severe (more than 30 events/hour).
Walking distance | Before and after intervention (12 weeks)
  The six-minute walking test (6MWT) will be used to determine walking distance, in meters (m), covered during six minutes. A 20-meter indoor corridor will be used and patients will be encouraged to walk as much as possible during that time.
1-minute Sit-to-Stand test | Before and after intervention (12 weeks)
  Number of sit-to- stand repetitions done in 1 minute (STS-1m). A 46-cm high chair will be used.

SECONDARY OUTCOMES:
Sleep quality | Before and after intervention (12 weeks)
  The Pittsburgh sleep quality index (PSQI) assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce 2one global score. The PSQI questions are rated from 0 = no difficulty to 3 = severe difficulty, generating scores that correspond to the domains of the scale. The scores range from 0 to 21 and a score >5 be considered as a significant sleep disturbance.
Resting heart rate | Before and after intervention (12 weeks)
  Number of beats in which you pump the least amount of blood necessary, because you are not doing physical activity. This is measured in the number of beats per minute taken at complete rest.
Blood pressure | Before and after intervention (12 weeks)
  It´s the pressure of circulating blood against the walls of blood vessels. Blood pressure is usually expressed in terms of the systolic pressure (maximum pressure during one heartbeat) over diastolic pressure (minimum pressure between two heartbeats) in the cardiac cycle. It is measured in millimetres of mercury (mmHg) above the surrounding atmospheric pressure, or in kilopascals (kPa).
Glycosylated hemoglobin | Before and after intervention (12 weeks)
  It´s a blood test that measures the average blood glucose level over the past two to three months, showing the percentage of hemoglobin (the protein that carries oxygen) that has been coated with sugar. Non-diabetic level: ≤ 5.6%; in practice it rules out the diagnosis of diabetes; Prediabetic level (increased risk of diabetes or prediabetes): between 5.7% and 6.4%; Diabetic level: ≥ 6.5%, which is compatible with the diagnosis of diabetes.
Lipid Profile | Before and after intervention (12 weeks)
  A lipid profile is a blood test to measure different types of lipids, this is used to determine lipid metabolism as well as the risk of developing cardiovascular pathologies. These include total cholesterol and triglycerides, which are measured in milligrams per deciliter (mg/dL).
Body composition | Before and after intervention (12 weeks)
  BIA (Bioelectrical Impedance) body composition is a noninvasive method that assesses the distribution of fat, muscle, and water in the body by sending a low-intensity electrical current through the tissues and measuring the resistance it offers. Comprehensive body composition analysis measures 9 key metrics including weight, body fat, muscle mass, body water percentage, bone mass and visceral fat.
Health-related quality of life | Before and after intervention (12 weeks)
  Component of quality of life in general that is due to the health care conditions of people and that is referred to from the subjective experiences of patients about their global health. The SF-36 Health Questionnaire is a 36-question instrument used to assess health-related quality of life, from the patient's perspective. It consists of eight scales that measure different aspects of health, such as physical function, physical role, bodily pain, general health, vitality, social function, emotional role, and mental health. Responses are coded and recoded, and results are converted to a scale from 0 to 100, with 0 representing the worst health and 100 the best.
Anxiety and depression | Before and after intervention (12 weeks)
  The "HAD questionnaire" refers to the Hospital Anxiety and Depression Scale (HADS), a 14-item questionnaire used to assess emotional distress in patients, particularly those with physical illnesses. It consists of two subscales, one for anxiety and one for depression, which are scored separately to identify the severity of both problems. The total score for each subscale (anxiety and depression) ranges from 0 to 21. Interpretation of results: Anxiety and Depression Subscale: (0-7): Absence of symptoms. (8-10): Doubtful symptoms. (11) or more: Certain symptoms.
Risk of developing obstructive sleep apnea | Before and after intervention (12 weeks)
  The STOP-Bang scale is a simple and widely used screening questionnaire to assess the risk of developing obstructive sleep apnea (OSA).
  The questionnaire consists of eight "Yes" or "No" answer questions, divided into two groups that give the scale its name: Snoring, Tired, Observed, Pressure, Body mass index, Age, Neck and Gender. Interpretation of the score:
  Low risk of OSA: 0 to 2 affirmative answers. Intermediate risk of OSA: 3 to 4 affirmative answers. High risk of OSA: 5 or more affirmative answers, or if specific criteria are met, such as answering "Yes" to 2 or more STOP questions plus a large neck circumference or male gender.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Vilaro, Phd, Study Chair — University Ramon Llull
Locations (1):
- Carlos Andrade Marín Hospital, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: No